CLINICAL TRIAL: NCT04991831
Title: A Post-Approval Registry for Exablate 4000 Type 1.0 and Type 1.1 for Unilateral Thalamotomy for the Treatment of Medication-Refractory Tremor Dominant Idiopathic Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Other Study IDs: PD012
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Tremor Associated With Tremor Dominant Parkinson's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post Exablate Neuro Thalamotomy for Tremor Associated with Tremor Dominant Parkinson's Disease: This is a post Exablate Neuro Thalamotomy registry. No intervention is performed under this registry protocol.
  Interventions: Device: Unilateral thalamotomy

INTERVENTIONS:
Device: Unilateral thalamotomy — Unilateral thalamotomy using focused ultrasound for the treatment of medication-refractory tremor dominant idiopathic Parkinson's Disease.

SUMMARY:
The objectives of this study are to collect the long-term safety and effectiveness data of performing thalamotomy for tremor dominant Parkinson's Disease (TDPD) using the Exablate Neuro system.

DETAILED DESCRIPTION:
This is a post-approval registry which is required by of the approval under PMA P150038/S006 for the Exablate® Model 4000 (Exablate Neuro) Type 1.0 and Type 1.1 for unilateral thalamotomy in the treatment of medication refractory Tremor Dominant Parkinson's Disease (TDPD). Subjects participating in this registry will have received a unilateral thalamotomy (ventralis medius) prior to enrollment using the commercially available Exablate Neuro for the treatment of Essential tremor and TDPD.

The following assessments will be collected at Baseline,1, 3, 6, and 12 months post Exablate procedure and annually thereafter for 5 years:

* Adverse Events (AEs) (does not apply to Baseline Visit)
* Medication usage
* Clinical Rating Scale for Tremor (CRST) ON medication
* Unified Parkinson's Disease Rating Scale Part III ON medication
* EQ-5D-5L
* WPAI-GH

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subject undergoing an Exablate procedure for their planned TDPD treatment; per local institution standard of care.
3. Subject is willing to cooperate with the Registry requirements including compliance with the regimen and completion of all study visits
4. Subject has signed and received a copy of the approved informed consent form

Exclusion Criteria:

Subject does not agree to participate or is unlikely to participate for the entirety of the study.

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population enrolled in this registry will be comprised of male and female patients that plan to be treated for TDPD using the Exablate Neuro system.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Long-term adverse events. | Five years.
  This registry will collect the long-term safety data after performing thalamotomy for TDPD using the Exablate Neuro system.

SECONDARY OUTCOMES:
Tremor/motor intensity and impact on disability | Five years.
  Long term tremor motor scores and the impact of tremor on disability will be monitored using components of the Clinical Rating Scale for Tremor (CRST)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Miami Neuroscience Institute Baptist Health, Miami, Florida
  - Rush University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Novant Health Brain & Spine Surgery, Huntsville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Fairborn, Ohio
- University of Dundee, Dundee, Scotland, United Kingdom